CLINICAL TRIAL: NCT00401843
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study Comparing the Combination of CNTO 328 (Anti-IL-6 Monoclonal Antibody) and Velcade Versus Velcade Alone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of the Safety and Efficacy of CNTO 328 and Bortezomib to Bortezomib Alone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012784; C0328T06 (Other: Janssen Research & Development, LLC); 2006-001904-36 (EudraCT Number)
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Monoclonal Antibody; Intravenous; refractory or relapsed multiple myeloma; velcade; bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — siltuximab; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Device: No

ARMS (3):
- Part 1: Siltuximab Plus Bortezomib (Experimental): Siltuximab 6 milligram per kilogram (mg/kg) will be administered as intravenous infusion once every 2 weeks along with bortezomib 1.3 milligram per square meter (mg/m^2) during cycle 1.
  Interventions: Biological: Siltuximab; Drug: Bortezomib
- Part 2: Bortezomib + Placebo (Experimental): Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 4, 8, 11, followed by a 10-day rest period; and on Days 22, 25, 29, and 32 followed by a 10-day rest period along with matching placebo administered as intravenous infusion once every 2 weeks during 42-day treatment phase. Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 8, 15, 22 followed by a 13-day rest period (cycle Days 23 to 35) along with matching placebo once every 2 weeks during 35-day Maintenance Phase. Dexamethasone tablet will be administered at first occurrence of documented disease progression or if bortezomib was discontinued due to intolerable toxicity. Dexamethasone 40 milligram per day (mg/day) will be administered on days 1-4, 9-12, and 17-20 for four 28-day cycles then 40 mg/day for Days 1-4 for all subsequent cycles.
  Interventions: Drug: Bortezomib; Drug: Placebo; Drug: Dexamethasone
- Part 2: Bortezomib + Siltuximab (Experimental): Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 4, 8, 11, followed by a 10-day rest period; and on Days 22, 25, 29, and 32 followed by a 10-day rest period along with Siltuximab administered as intravenous infusion once every 2 weeks during 42-day treatment phase. Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 8, 15, 22 followed by a 13-day rest period (cycle Days 23 to 35) along with Siltuximab administered as intravenous infusion once every 2 weeks for 35-day Maintenance Phase. Dexamethasone tablet will be administered at first occurrence of documented disease progression or if bortezomib was discontinued due to intolerable toxicity. Dexamethasone 40 mg/day will be administered on days 1-4, 9-12, and 17-20 for four 28-day cycles then 40 mg/day for Days 1-4 for all subsequent cycles.
  Interventions: Biological: Siltuximab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Biological: Siltuximab — Siltuximab 6 mg/kg will be administered as intravenous infusion once every 2 weeks during cycle 1 in Part 1. Siltuximab 6 mg/kg will be administered as intravenous infusion once every 2 weeks during 42-day Treatment Phase and 35-day Maintenance Phase in Part 2.
  Other Names: CNTO 328
  Arms: Part 1: Siltuximab Plus Bortezomib; Part 2: Bortezomib + Siltuximab
Drug: Bortezomib — Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus once every 2 weeks during cycle 1 in Part 1. Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 4, 8, 11, followed by a 10-day rest period; and on Days 22, 25, 29, and 32 followed by a 10-day rest period during 42-day treatment phase in Part 2. Bortezomib 1.3 mg/m2 will be administered as intravenous bolus on Days 1, 8, 15, 22 followed by a 13-day rest period (cycle Days 23 to 35) during 35-day Maintenance Phase in Part 2.
  Other Names: VELCADE
Drug: Placebo — Matching placebo will be administered as intravenous infusion once every 2 weeks during 42-day treatment phase and 35-day maintenance phase in Part 2.
  Arms: Part 2: Bortezomib + Placebo
Drug: Dexamethasone — Dexamethasone tablet will be administered in this study at the first occurrence of documented disease progression or if bortezomib was discontinued due to intolerable toxicity. Dexamethasone 40 mg/day will be administered on days 1-4, 9-12, and 17-20 for four 28-day cycles then 40 mg/day for Days 1-4 for all subsequent cycles in treatment phase and maintenance phase of Part 2.
  Arms: Part 2: Bortezomib + Placebo; Part 2: Bortezomib + Siltuximab

SUMMARY:
The purpose of Part 1 of the study is to determine the safety of the combination of Siltuximab (CNTO 328) and bortezomib (Velcade). The purpose of Part 2 of the study is to compare the length of progression free survival for those patients given CNTO 328 and bortezomib to those patients given bortezomib alone.

DETAILED DESCRIPTION:
The purpose of this study is to see what effects CNTO 328 has on relapsed or refractory multiple myeloma. The study drug, CNTO 328, is a chimeric (part mouse) antibody (small protein that is important for fighting infection).CNTO 328 blocks a small protein called Interleukin 6 (IL-6). IL-6 is made naturally by your body, and at normal levels is important for inflammatory response. High levels of IL-6 can help cancer cells grow and interfere with chemotherapy drugs killing cancer cells. Cancer-related sickness such as cachexia (weight loss), bone resorption (weakening of your bones), and depression have been linked to high levels of IL-6. CNTO 328 has been shown to slow down tumor growth or shrink tumors when tested in animals. In other clinical trials, over 100 patients have received CNTO 328. There are studies ongoing in participants with kidney cancer, hematologic malignancies (blood cancers such as multiple myeloma), and prostate cancer, to see if CNTO 328 is safe and to see what effects it has on these types of cancer. At this time, it is unknown what effect CNTO 328 has had on the participants' cancer. Bortezomib is a type of drug known as a "proteasome inhibitor." A proteasome is a substance that is found in every cell and it is there to help to break down other substances ('proteins') and has a role in the way cells divide. If the proteasome is inhibited, it cannot perform its function in the cell, and if a cell cannot divide it dies. Over 8000 patients with multiple myeloma and other types of cancer have been treated with bortezomib. Bortezomib has been extensively studied in patients with previously treated multiple myeloma. Based on its established activity in pretreated multiple myeloma, bortezomib is registered in the United States and in Europe for the treatment of multiple myeloma patients who have received at least two prior therapies and have demonstrated disease progression on the last therapy. Bortezomib is currently also being studied in several other cancer types.This study consists of two parts. The purpose of Part 1 is to determine the safety of CNTO 328 and bortezomib when given together as a treatment. The purpose of Part 2 is to compare the safety and effects (good and bad) of the combination of CNTO 328 and bortezomib to the safety and effects of bortezomib alone. About 20 patients will take part in the first part of the study. About 270 patients will take part in the second part of the study at approximately 70 sites in the US, Canada, and Europe. Patients will be in the study for about 12 months, with a follow-up period of around 9 months. The study is divided into four different phases: Screening phase-which lasts up to 4 weeks. During this phase the study doctor will perform tests to see if the patient can participate in the study.Treatment phase-which may last up to 4 cycles of 42 days each during which the patient will be treated with CNTO 328 and bortezomib. Maintenance phase-If the patient benefits from the therapy in the treatment phase, the patient will continue to receive CNTO 328 and bortezomib, but now in cycles of 35 days each. Follow up phase, this includes an end of treatment visit 4 weeks after the patient's last infusion and follow up visits every three months until the patient starts a new anti-cancer treatment. CNTO 328 6mg/kg ( 6 milligrams per kilogram of body weight) will be given intravenously (into the vein) over 2 hours once every 2 weeks. Patients who respond with stable disease or better may receive additional doses. Bortezomib will be given IV (into the vein) at 1.3 mg/m2 over 3-5 seconds twice a week for 2 weeks followed by 1 week of rest.

ELIGIBILITY:
Inclusion Criteria:

* Measurable secretory disease defined as either serum monoclonal paraprotein, (M-protein) greater than or equal to (>=)1 gram per deciliter (g/dL) or urine monoclonal (light chain) protein (> 200 mg/24 hours)
* Documented disease progression after at least 1 prior line of therapy but no more than 3 or have had no response to previous treatment (primary refractory disease)
* ECOG performance status score of less than or equal to (<=) 2
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* No prior treatment with bortezomib
* Not Refractory to high-dose dexamethasone
* Not >= Grade 2 peripheral neuropathy
* Have not received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant
* No prior or concomitant malignancy (other than multiple myeloma) except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or other cancer for which the patient has been disease-free for <= 3 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2006-11-28 (Actual); Primary Completion 2011-08-16 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (80):
- United States (11):
  - Greenbrae, California
  - Los Angeles, California
  - Indianapolis, Indiana
  - Albuquerque, New Mexico
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - North Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Madison, Wisconsin
- Belgium (5):
  - Antwerp
  - B-8000 Brugge
  - Brussels
  - Edegem
  - Leuven
- Rio de Janeiro, Brazil
- Bulgaria (3):
  - Bulgaria
  - Pleven
  - Plovdiv
- Canada (3):
  - Vancouver, British Columbia
  - Québec, Quebec
  - Calgary
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- France (5):
  - Grenoble
  - Lille Cedex N/a
  - Montpellier
  - Pierre-Bénite
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Aschaffenburg
  - Essen
  - Mainz
  - Münster
  - Stuttgart
  - Ulm
- Athens, Greece
- Hungary (5):
  - Budapest
  - Debrecen
  - Gyõr
  - Nyíregyháza
  - Szeged
- Netherlands (4):
  - Amersfoort
  - Amsterdam
  - Rotterdam
  - The Hague
- Poland (7):
  - Bialystok
  - Gdansk
  - Katowice
  - Lodz
  - Lublin
  - Poznan
  - Wroclaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Romania (5):
  - Baia Mare
  - Brasov
  - Bucharest
  - Iași
  - Tg Mures
- Russia (7):
  - Arkhangelsk
  - Izhevsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Ufa
- Slovakia (2):
  - Bratislava
  - Martin
- Spain (5):
  - Badalona
  - Barcelona
  - Madrid
  - Salamanca
  - Valencia
- United Kingdom (4):
  - London
  - Nottingham
  - Plymouth
  - Sutton

REFERENCES:
- [Derived] Orlowski RZ, Gercheva L, Williams C, Sutherland H, Robak T, Masszi T, Goranova-Marinova V, Dimopoulos MA, Cavenagh JD, Spicka I, Maiolino A, Suvorov A, Blade J, Samoylova O, Puchalski TA, Reddy M, Bandekar R, van de Velde H, Xie H, Rossi JF. A phase 2, randomized, double-blind, placebo-controlled study of siltuximab (anti-IL-6 mAb) and bortezomib versus bortezomib alone in patients with relapsed or refractory multiple myeloma. Am J Hematol. 2015 Jan;90(1):42-9. doi: 10.1002/ajh.23868. PMID 25294016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 144 participants were randomized to bortezomib plus placebo group; of which, 3 participants received incorrect treatment (bortezomib plus siltuximab).
Groups:
- Part 1 - Bortezomib + Siltuximab: Siltuximab 6 milligram per kilogram (mg/kg) will be administered as intravenous infusion once every 2 weeks along with bortezomib 1.3 milligram per square meter (mg/m^2) during cycle 1.
- Part 2 - Bortezomib + Placebo: Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 4, 8, 11, followed by a 10- day rest period; and on Days 22, 25, 29, and 32 followed by a 10-day rest period along with matching placebo administered as intravenous infusion once every 2 weeks during 42-day treatment phase.
  Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 8, 15, 22 followed by a 13- day rest period (cycle Days 23 to 35) along with matching placebo once every 2 weeks during 35-day Maintenance Phase. Dexamethasone tablet will be administered at first occurrence of documented disease progression or if bortezomib was discontinued due to intolerable toxicity. Dexamethasone 40 milligram per day (mg/day) will be administered on days 1-4, 9-12, and 17-20 for four 28-day cycles then 40 mg/day for Days 1-4 for all subsequent cycles.
- Part 2 - Bortezomib + Siltuximab: Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 4, 8, 11, followed by a 10- day rest period; and on Days 22, 25, 29, and 32 followed by a 10-day rest period along with Siltuximab administered as intravenous infusion once every 2 weeks during 42-day treatment phase. Bortezomib 1.3 mg/m^2 will be administered as intravenous bolus on Days 1, 8, 15, 22 followed by a 13-day rest period (cycle Days 23 to 35) along with Siltuximab administered as intravenous infusion once every 2 weeks for 35-day Maintenance Phase. Dexamethasone tablet will be administered at first occurrence of documented disease progression or if bortezomib was discontinued due to intolerable toxicity.
  Dexamethasone 40 mg/day will be administered on days 1-4, 9-12, and 17-20 for four 28-day cycles then 40 mg/day for Days 1-4 for all subsequent cycles.
Period: Overall Study
Arm/Group | Part 1 - Bortezomib + Siltuximab | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Started | 21 | 144 | 142
Treated | 21 | 142 | 139
Completed | 0 | 0 | 0
Not Completed | 21 | 144 | 142
Not completed — Achieved Complete Response | 1 | 5 | 11
Not completed — Adverse Event | 7 | 26 | 27
Not completed — Death | 0 | 8 | 10
Not completed — Disease progression | 10 | 60 | 49
Not completed — End of Study | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Other Unspecified | 0 | 3 | 5
Not completed — Physician Decision | 0 | 16 | 10
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 5
Not completed — Withdrawal of consent to study agent | 1 | 15 | 17
Not completed — Randomized but not Treated | 0 | 2 | 3
Not completed — Received incorrect treatment | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Bortezomib + Siltuximab | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab | Total
Number analyzed (Participants) | 21 | 144 | 142 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.76) | 62.3 (9.65) | 63.5 (9.32) | 63.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 59 | 70 | 142
  Male | 8 | 85 | 72 | 165
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 2 | 1 | 3
  Brazil | 0 | 6 | 4 | 10
  Bulgaria | 0 | 16 | 10 | 26
  Canada | 3 | 4 | 5 | 12
  Czech Republic | 0 | 13 | 11 | 24
  France | 7 | 5 | 7 | 19
  Germany | 0 | 1 | 1 | 2
  Greece | 0 | 5 | 5 | 10
  Hungary | 0 | 10 | 10 | 20
  Netherlands | 2 | 4 | 5 | 11
  Poland | 0 | 19 | 11 | 30
  Portugal | 0 | 5 | 4 | 9
  Romania | 0 | 8 | 5 | 13
  Russian Federation | 0 | 21 | 27 | 48
  Spain | 2 | 5 | 10 | 17
  United Kingdom | 0 | 12 | 15 | 27
  United States | 7 | 8 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time interval between randomization and the first documented sign of disease progression (including relapse from complete response [CR]) by the European Bone Marrow Transplant (EBMT) criteria or death, whichever occurred first. Relapse from CR requires at least 1 of the following: Reappearance of serum or urinary M-protein on immunofixation or routine electrophoresis, confirmed by at least 1 further investigation and excluding oligoclonal immune reconstitution; Greater than or equal to (>=) 5 percent (%) plasma cells either in a bone marrow aspirate or on trephine bone biopsy; Development of new lytic bone lesions or soft tissue plasmacytomas or definite increase in the size of residual bone lesions (development of a compression fracture does not exclude continued response and may not indicate progression); Development of hypercalcemia not attributable to any other cause.
Time Frame: Randomization until disease progression or death, which ever occured first (maximum up to 5 years)
Population: Intent-to-treat (ITT) population included all participants randomized in Part 2. Participants were analyzed as per initial randomization.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Number analyzed (Participants) | 144 | 142
days | 232 [191 to 302] | 245 [217 to 300]

2. Secondary Outcome: Percentage of Participants With Best Confirmed Response of Complete Response (CR) or Partial Response (PR) (Overall Response Rate)
Description: Overall response rate was defined as best response (CR/PR confirmed) for a participant recorded from first administration of study agent or randomization (Part 2) until disease progression/recurrence and before dexamethasone was added. CR: Absence of original M-protein in serum/urine by immunofixation,maintained for minimum of 6 weeks. The presence of oligoclonal bands consistent with oligoclonal immune reconstitution does not exclude CR; Less than 5 percent (%) plasma cells in bone marrow aspirate and also on trephine bone biopsy if biopsy is performed; No increase in size/number of lytic bone lesions; Disappearance of soft tissue plasmacytomas. PR: Greater than or equal to (>=) 50% reduction in level of serum M-protein, maintained for minimum of 6 weeks. Reduction in 24 hour urinary light chain excretion either by >= 90% or to < 200 mg, maintained for minimum of 6 weeks; >= 50% reduction in size of soft tissue plasmacytomas; No increase in size/number of lytic bone lesions.
Time Frame: Randomization until disease progression (maximum up to 5 years)
Population: Response-evaluable population:all participants in Part 2 with confirmed diagnosis of multiple myeloma and measurable,secretory disease:either serum M-protein 1 >= gram per deciliter(g/dL)/urine M-protein >200 mg per 24 hours,at study entry;had at least 1 study agent administration;at least 1 post-baseline disease assessment before dexamethasone.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Number analyzed (Participants) | 137 | 131
percentage of participants | 46.7 | 55.0

3. Secondary Outcome: Percentage of Participants With Confirmed Complete Response (CR Rate)
Description: CR rate was defined as the percentage of participants who achieved a confirmed CR before dexamethasone was added. CR: Absence of original M-protein in serum/urine by immunofixation,maintained for minimum of 6 weeks. The presence of oligoclonal bands consistent with oligoclonal immune reconstitution does not exclude CR; Less than 5 percent (%) plasma cells in bone marrow aspirate and also on trephine bone biopsy if biopsy is performed; No increase in size/number of lytic bone lesions; Disappearance of soft tissue plasmacytomas.
Time Frame: Randomization until disease progression (maximum up to 5 years)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Number analyzed (Participants) | 137 | 131
percentage of participants | 7.3 | 10.7

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the first administration of study agent or randomization (Part 2) and the participant's death from any cause. For participants with unknown survival status as of the data cut-off date, overall survival was censored at the last date known to be alive.
Time Frame: up to 5 years
Population: ITT population included all participants randomized in Part 2. Participants were analyzed as per initial randomization.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Number analyzed (Participants) | 144 | 142
days | 1121 [1038.0 to NA] — Upper limit of 95% CI was not estimable due to high censorship rate and lesser number of events. | 937 [713 to 1127]

5. Primary Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: up to 5 years
Population: The safety population included all participants who received at least 1 dose of study treatment in Part 1 or Part 2. Participants were analyzed as per actual treatment received.
Measure: Number; unit: participants
Arm/Group | Part 1 - Bortezomib + Siltuximab | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Number analyzed (Participants) | 21 | 139 | 142
participants
  Adverse Events (AEs) | 21 | 138 | 140
  Serious Adverse Events (SAEs) | 10 | 44 | 47

ADVERSE EVENTS:
Description: The safety population included all participants who received at least 1 dose of study treatment in Part 1 or Part 2. Participants were analyzed as per actual treatment received.
Arm/Group | Part 1 - Bortezomib + Siltuximab | Part 2 - Bortezomib + Placebo | Part 2 - Bortezomib + Siltuximab
Serious Adverse Events (participants affected / at risk) | 10/21 | 44/139 | 47/142
Other Adverse Events (participants affected / at risk) | 21/21 | 135/139 | 140/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Bortezomib + Siltuximab (N=21) | Part 2 - Bortezomib + Placebo (N=139) | Part 2 - Bortezomib + Siltuximab (N=142)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac Disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 1
Eye Swelling (Eye disorders) | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 1
Chills (General disorders) | 0 | 1 | 0
Chronic Fatigue Syndrome (General disorders) | 0 | 0 | 1
Face Oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1 | 0
Mass (General disorders) | 1 | 0 | 0
Performance Status Decreased (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Sudden Cardiac Death (General disorders) | 0 | 0 | 1
Sudden Death (General disorders) | 0 | 2 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Acute Hepatitis B (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 3 | 2
Endocarditis (Infections and infestations) | 0 | 0 | 1
Enterobacter Bacteraemia (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 1 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 2 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Meningitis Bacterial (Infections and infestations) | 0 | 0 | 1
Meningitis Pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 6 | 5
Pneumonia Pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia Streptococcal (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 4
Septic Shock (Infections and infestations) | 0 | 1 | 0
Streptococcal Bacteraemia (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2
Varicella (Infections and infestations) | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone Lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1
Mononeuritis (Nervous system disorders) | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2
Viith Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0
Vocal Cord Paresis (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Obstructive Uropathy (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 1 | 2
Renal Failure Acute (Renal and urinary disorders) | 1 | 1 | 3
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Mediastinal Shift (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Bortezomib + Siltuximab (N=21) | Part 2 - Bortezomib + Placebo (N=139) | Part 2 - Bortezomib + Siltuximab (N=142)
Anaemia (Blood and lymphatic system disorders) | 9 | 46 | 45
Leukopenia (Blood and lymphatic system disorders) | 8 | 16 | 38
Lymphopenia (Blood and lymphatic system disorders) | 8 | 5 | 13
Neutropenia (Blood and lymphatic system disorders) | 17 | 53 | 86
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 65 | 83
Vertigo (Ear and labyrinth disorders) | 2 | 6 | 6
Chalazion (Eye disorders) | 2 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 5 | 7
Lacrimation Increased (Eye disorders) | 2 | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 3 | 10 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 8 | 7
Aphthous Stomatitis (Gastrointestinal disorders) | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 12 | 22 | 31
Diarrhoea (Gastrointestinal disorders) | 13 | 50 | 53
Dyspepsia (Gastrointestinal disorders) | 3 | 9 | 13
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 42 | 40
Stomatitis (Gastrointestinal disorders) | 3 | 4 | 6
Vomiting (Gastrointestinal disorders) | 4 | 28 | 28
Asthenia (General disorders) | 5 | 27 | 24
Chills (General disorders) | 3 | 6 | 6
Fatigue (General disorders) | 8 | 40 | 39
Gait Disturbance (General disorders) | 2 | 1 | 1
Influenza Like Illness (General disorders) | 3 | 5 | 4
Oedema Peripheral (General disorders) | 4 | 16 | 16
Pyrexia (General disorders) | 3 | 27 | 8
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 14 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 5
Bronchitis (Infections and infestations) | 3 | 11 | 14
Ear Infection (Infections and infestations) | 2 | 0 | 1
Herpes Simplex (Infections and infestations) | 2 | 2 | 4
Herpes Zoster (Infections and infestations) | 2 | 13 | 4
Hordeolum (Infections and infestations) | 3 | 2 | 6
Nasopharyngitis (Infections and infestations) | 3 | 13 | 15
Pneumonia (Infections and infestations) | 3 | 4 | 7
Respiratory Tract Infection (Infections and infestations) | 2 | 11 | 14
Rhinitis (Infections and infestations) | 1 | 7 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 12 | 14
Urinary Tract Infection (Infections and infestations) | 3 | 7 | 12
Weight Decreased (Investigations) | 7 | 20 | 20
Weight Increased (Investigations) | 3 | 3 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 28 | 32
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 6
Enzyme Abnormality (Metabolism and nutrition disorders) | 1 | 9 | 5
Hyperamylasaemia (Metabolism and nutrition disorders) | 3 | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 8 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 9
Hyperlipasaemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 6 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 7 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 13 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 9 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 19 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 17 | 23
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 29 | 21
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 15 | 17
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 11
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 10 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 12
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 15 | 25
Balance Disorder (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 10 | 14
Dysgeusia (Nervous system disorders) | 2 | 2 | 4
Headache (Nervous system disorders) | 8 | 14 | 18
Hypoaesthesia (Nervous system disorders) | 0 | 7 | 5
Lethargy (Nervous system disorders) | 0 | 7 | 7
Neuralgia (Nervous system disorders) | 1 | 33 | 31
Paraesthesia (Nervous system disorders) | 3 | 16 | 14
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 8 | 8
Peripheral Sensory Neuropathy (Nervous system disorders) | 9 | 73 | 73
Anxiety (Psychiatric disorders) | 4 | 6 | 8
Insomnia (Psychiatric disorders) | 5 | 15 | 15
Renal Failure (Renal and urinary disorders) | 2 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 2 | 4 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 18 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 14 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 14 | 15
Haematoma (Vascular disorders) | 2 | 1 | 2
Hypertension (Vascular disorders) | 4 | 9 | 18
Hypotension (Vascular disorders) | 4 | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.